CLINICAL TRIAL: NCT02653872
Title: An Open-label, Non-randomized, Fixed Sequence Study Assessing the Pharmacokinetics of AZD7986 When Administered Alone and With Multiple Doses of Verapamil and Itraconazole or Diltiazem in Healthy Subjects
Brief Title: A Phase I Study to Assess PK of AZD7986 Alone & With Verapamil, Itraconazole or Diltiazem in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D6190C00003
Record Dates: First submitted 2016-01-11; First posted 2016-01-12 (Estimated); Results first posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2017-07

CONDITIONS: Healthy Subjects
Keywords: Non-randomized; Verapamil; Itraconazole; Diltiazem; Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — brensocatib; Verapamil; Itraconazole; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD7986 (alone) Treatment period 1 (Experimental): AZD7986 (15 mg/mL) 25 mg dosage administered alone
  Interventions: Drug: AZD7986
- Verapamil (with AZD7986) Treatment period 2 (Active Comparator): Daily administration of verapamil (240 mg, extended release formulation) on Days 1 to 10 plus administration of single dose AZD7986 (25 mg) on Day 5
  Interventions: Drug: AZD7986; Drug: Verapamil
- Itraconazole (with AZD7986) Treatment Period 3 (Active Comparator): Itraconazole (200 mg, oral solution formulation 10 mg/mL) administered twice on Day 1 and then daily Days 2 to 11 plus single dose AZD7986 (25 mg, tbc) on Day 6
  Interventions: Drug: AZD7986; Drug: Itraconazole
- Diltiazem (with AZD7986) Treatment period 3 (Active Comparator): Diltiazem (360 mg, extended release formulation) administered Days 1 to 13 plus single dose AZD7986 (25 mg) on Day 8
  Interventions: Drug: AZD7986; Drug: Diltiazem

INTERVENTIONS:
Drug: AZD7986 — Oral solution, single dose, dilution from concentrate
Drug: Verapamil — Extended release tablet for oral use
  Arms: Verapamil (with AZD7986) Treatment period 2
Drug: Itraconazole — Oral solution
  Arms: Itraconazole (with AZD7986) Treatment Period 3
Drug: Diltiazem — Extended release capsule
  Arms: Diltiazem (with AZD7986) Treatment period 3

SUMMARY:
This is a phase 1, non-randomized, fixed sequence, 3-period, drug-drug interaction study to assess the pharmacokinetics (PK) of AZD7986 in healthy subjects when administered alone and in combination with multiple doses of verapamil and itraconazole or diltiazem

DETAILED DESCRIPTION:
This study will be an open-label, non-randomised, fixed sequence, 3-period study conducted at a single study centre to assess the PK of AZD7986 in healthy subjects when administered alone and in combination with multiple doses of verapamil and itraconazole or diltiazem. An adaptive design with an interim analysis of the PK data from Periods 1 and 2 will be used to determine which of itraconazole or diltiazem will be administered in combination with AZD7986 in Period 3.

Treatments to be administered in a fixed order separated by a washout period:

period 1 - single AZD7986 (25 mg) on Day 1 (1 hour before food), washout 7 days period 2 - verapamil (240 mg extended release formulation) daily 1 hour before food (Day 1 to 10) and a single dose of AZD7986 (25 mg) 1 hour before food (Day 5), washout period 14 days period 3 - subject to interim pharmacokinetic analysis of AZD7986 alone compared with AZD7986 and verapamil combined, either itraconazole (200 mg, oral solution formulation 10mg/mL) administered twice on Day 1 and daily on days 2 to 11 (1 hour before food) plus AZD7986 (25mg) single dose on Day 6 (1 hour before food); or diltiazem (360 mg, extended release formulation) on Days 1 to 13 (1 hour before food) plus AZD7986 (25 mg) 1 hour before food on Day 8.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venepuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post menopausal range(> 40 milli-International unit [mIU]/mL).

   Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive.
5. Provision of signed, written and dated informed consent for optional genetic/biomarker research.
6. Hormone replacement therapy is not allowed for females to exclude any drug drug interaction between the hormone replacement therapy and AZD7986.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of AZD7986.
4. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator.
5. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
6. Any clinically significant abnormal findings in vital signs after at least 10 minutes of rest, defined as the following:

   * Systolic blood pressure < 100 mmHg or > 140 mmHg;
   * Diastolic blood pressure < 50 mmHg or > 90 mmHg; or
   * Pulse rate < 50 or > 85 beats per minute.
7. Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 Lead ECG as considered by the investigator that may interfere with the interpretation of ECG interval measured from the onset of the QRS complex (electrical activity or ventricular contraction on the ECG where Q represents the downward deflection, R represents upward deflection and S represents a downward one) to the end of the T wave corrected for heart rate (QTc) interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
8. Prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.
9. PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
10. PR (PQ) interval prolongation > 200 ms, intermittent second or third degree atrioventricular (AV) block (Wenckebach block while asleep is not exclusive), or AV dissociation.
11. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
12. Known or suspected history of drug abuse, as judged by the investigator.
13. Current smokers or those who have smoked or used nicotine products within the 3 months before screening.
14. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the investigator.
15. Positive screen for drugs of abuse or cotinine at screening or on each admission to the study centre or positive screen for alcohol on each admission to the study unit.
16. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7986.
17. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the investigator.
18. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of AZD7986.
19. Use of any prescribed or non-prescribed medication including antacids and other drugs for gastric acid-related disorders, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of AZD7986 or longer if the medication has a long half-life.

    Note: Hormonal replacement therapy is not allowed for females.
20. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
21. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of AZD7986 in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.

    Note: Subjects consented and screened, but not dosed in this study or a previous phase I study, are not excluded.
22. Subjects who have previously received AZD7986.
23. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
24. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
25. Subjects who cannot communicate reliably with the investigator.
26. Subjects who are vegans or have medical dietary restrictions.
27. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
28. Subject has increased risk of infection:

    * History and/or presence of tuberculosis (TB); positive result for interferon gamma release assay (IGRA) (i.e., QuantiFERON TB-Gold), subjects who have resided in regions where tuberculosis and mycosis are endemic during 90 days before screening, or who intend to visit such a region during the duration of the study i.e., deserts areas, Eastern Europe, Central and South America, Africa except Egypt, Russia, Asia, Indonesia. The test may be repeated if the initial test result is indeterminate.
    * Oral body temperature of > 37.7°C on Day -1, or as judged by the investigator.
    * Blood neutrophil count < 1.7 x109/L (Screening and Day -1 morning sample).
    * Is in high risk-group for HIV infection within the last 6 months (i.e., men who have had unprotected sex with men, women who have had sex without a condom with men who have sex with men, people who have had sex without a condom with a person who has lived or travelled in Africa, people who inject drugs, people who have had sex without a condom with somebody who has injected drugs, people who have caught another sexually transmitted infection, people who have received a blood transfusion while in Africa, Eastern Europe, the countries of the former Soviet Union, Asia or Central and Southern America).
    * Other latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) within 90 days of screening, or history of skin abscesses within 90 days of screening.
    * Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to screening, as determined by the investigator.
    * Subjects with active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
    * Disease history suggesting abnormal immune function.
    * Subjects who have received live or live-attenuated vaccine in the 4 weeks prior to dosing.
    * High-sensitivity C-reactive protein above upper limit of laboratory reference range at screening and on Day -1.
29. Subjects with a history or signs of current gingivitis/periodontitis or a history or current hyperkeratosis of palms and soles will be excluded. (Due to the fact that many subjects lacking functional DPP1 enzyme have been described to have periodontitis and palmoplantar hyperkeratosis.)
30. Subjects with total urinary protein/urine creatinine ratio outside the normal range.
31. Drugs affecting CYP3A4 should be refrained from use for 3 weeks prior to study commencement and thereafter until study completion.

    In addition, the following is considered a criterion for the exclusion from the optional genetic component of the study:
32. History of bone marrow transplant
33. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.
34. Hypersensitivity to the verapamil or to any of the excipients.
35. History of serious cardiac events such as myocardial infarction.
36. History of sino-atrial block; sick sinus syndrome; chronic or uncompensated heart failure (including left ventricular heart failure).
37. History of atrial flutter, atrial fibrillation or Wolff-Parkinson-White syndrome.
38. Known hypersensitivity to diltiazem or to any of the excipients.
39. Known hypersensitivity to itraconazole or to any of the excipients.
40. Elevated or abnormal liver enzymes or active liver disease, or who have experienced liver toxicity with other drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, FFPM, Principal Investigator — Parexel
Locations (1):
- Research Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL Early Phase Clinical Unit - London
Pre-assignment Details: Fifteen healthy male subjects were enrolled in the study to assess the pharmacokinetics (PK) of AZD7986 when administered alone (Treatment Period 1) and in combination with multiple doses of verapamil (Treatment Period 2) and itraconazole (Treatment Period 3).
Groups:
- All Participants: All 15 participants who were enrolled in the study and who received at least a single dose of the study drug in three treatment periods in a fixed sequence and were separated by a washout period.
Period: Overall Study
Arm/Group | All Participants
Started | 15
Treatment Period 1: | 15 (Participants received single AZD7986 (25 mg).)
Treatment Period 2: | 15 (Participants received Verapamil (240 mg; extended release formulation) + AZD7986 (25 mg).)
Treatment Period 3: | 15 (Participants received: itraconazole 200 mg + AZD7986.)
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fifteen participants were enrolled in this study. All participants signed and dated the informed consent document before any tests/procedures were performed. Of the 15 participants enrolled, all 15 were dosed and completed treatment. No participants were withdrawn during the study.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Effect of Verapamil and the Effect of Itraconazole on the PK of AZD7986 by Assessment of the Observed Maximum Plasma Concentration (Cmax).
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: Period 1,2&3: Day1 (AZD7986),Day5 (AZD7986+Verapamil) & Day6 (AZD7986): pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,5,8,9,12,24,48,72,96,120 & 144 hours post-dose; Period 3: Day6 (Itraconazole): pre-dose,0.25,0.5,0.75,1,1.5,2,3,4,5,8,9,12 & 24 hours post-dose
Population: The PK analysis set consisted of all subjects in the safety analysis set who received at least 1 dose of AZD7986 and for whom at least 1 of the primary PK parameters for AZD7986 could be calculated for at least 1 treatment period, and who had no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- AZD7986: Participants received a single dose of AZD7986 (25 mg) administration on Day 1 (1 hour before food).
- AZD7986 + Verapamil: Participants received Verapamil (240 mg; extended release formulation) administered daily (1 hour before food) on Days 1 to 10 plus administration of a single dose of AZD7986 (25 mg) on Day 5 (1 hour before food).
- AZD7986 + Itraconazole: Participants received Itraconazole (200 mg; oral solution formulation 10 mg/mL) administered twice on Day 1 and then daily on Days 2 to 11 (1 hour before food) plus administration of AZD7986 (25 mg) as a single dose on Day 6 (1 hour before food).
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
nmol/L | 385.8 (27.4) | 591.9 (27.1) | 234.1 (39.0)
Statistical Analysis 1: Comparison: AZD7986 vs AZD7986 + Verapamil; The study was designed based on a test for bioequivalence. Using an estimated standard deviation for Cmax of AZD7986 of less than or equal to 0.202, 12 evaluable subjects were deemed needed to achieve a power of 90%, at an assumed ratio of 0.95, to show that a two-sided 90% confidence interval for the ratio of Cmax between 2 treatments (AZD7986 and AZD7986+ Verapamil/Itraconazole) would be contained within the (0.8;1.25) equivalence limit. 3 extra subjects were added to compensate for dropout; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of Cmax for AZD7986 administered with verapamil over Cmax for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 153.40, 90% CI 2-sided [136.16 to 172.83]
Statistical Analysis 2: Comparison: AZD7986 vs AZD7986 + Itraconazole; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of Cmax for AZD7986 administered with itraconazole over Cmax for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 60.66, 90% CI 2-sided [53.84 to 68.34]

2. Primary Outcome: Effect of Verapamil and the Effect of Itraconazole on the PK of AZD7986 by Assessment of the Area Under Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC).
Description: To assess the effect of verapamil and itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
h*nmol/L | 6697 (44.8) | 8857 (43.3) | 7615 (35.1)
Statistical Analysis 1: Comparison: AZD7986 vs AZD7986 + Verapamil; The study was sized for Cmax primarily and not AUC. A two-sided 90% confidence interval for the ratio of AUC between the two treatments groups was used to determine equivalence; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of AUC for AZD7986 administered with verapamil over AUC for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 132.25, 90% CI 2-sided [121.78 to 143.64]
Statistical Analysis 2: Comparison: AZD7986 vs AZD7986 + Itraconazole; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of AUC for AZD7986 administered with itraconazole over AUC for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 113.70, 90% CI 2-sided [104.69 to 123.49]

3. Primary Outcome: Pharmacokinetics (PK) of AZD7986 by Assessment of the Area Under Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC [0-t]).
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
h*nmol/L | 6545 (44.8) | 8739 (43.5) | 7361 (34.4)
Statistical Analysis 1: Comparison: AZD7986 vs AZD7986 + Verapamil; The study was sized for Cmax primarily and not AUC (0-t). A two-sided 90% confidence interval for the ratio of AUC (0-t) between the two treatments groups was used to determine equivalence; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of AUC (0-t) for AZD7986 administered with verapamil over AUC (0-t) for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 133.51, 90% CI 2-sided [122.70 to 145.29]
Statistical Analysis 2: Comparison: AZD7986 vs AZD7986 + Itraconazole; [analysis description as in outcome 3, analysis 1]; Test type: Non-Inferiority or Equivalence — Geometric mean ratio of AUC (0-t) for AZD7986 administered with itraconazole over AUC (0-t) for AZD7986 administered alone. Presented as a percentage; ANOVA; % Geometric Mean Ratio = 112.45, 90% CI 2-sided [103.34 to 122.37]

4. Primary Outcome: Pharmacokinetics (PK) of AZD7986 by Assessment of Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t½λz).
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
hours | 23.35 (5.731) | 20.36 (4.812) | 27.89 (5.407)

5. Primary Outcome: Pharmacokinetics (PK) of AZD7986 by Assessment of the Time to Reach Maximum Plasma Concentration (Tmax)
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
hours | 0.75 [0.48 to 3.00] | 1.50 [0.73 to 1.52] | 1.50 [0.75 to 2.00]

6. Primary Outcome: Pharmacokinetics (PK) of AZD7986 by Assessment of the Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC (CL/F).
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
L/h | 9.807 (5.267) | 7.359 (3.765) | 8.308 (3.452)

7. Primary Outcome: Pharmacokinetics (PK) of AZD7986 by Assessment of the Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F).
Description: To assess the effect of Verapamil and Itraconazole on the PK of AZD7986.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole
Number analyzed (Participants) | 15 | 15 | 15
Litres | 297.1 (83.48) | 194.6 (41.68) | 317.8 (89.06)

8. Primary Outcome: Assessment of the Area Under the Plasma Concentration-curve Over the Dosing Interval (AUC [0 - τ]) of Verapamil, Itraconazole and OH-itraconazole Following Co-administration of AZD7986 With Verapamil or Itraconazole.
Description: To assess the area under the plasma concentration-time curve from time over the dosing interval tau (24 hours) of Verapamil, itraconazole and OH-itraconazole (a metabolite of Itraconazole) following co-administration of AZD7986 with Verapamil or Itraconazole.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Groups:
- Verapamil: Participants received Verapamil (240 mg; extended release formulation) administered daily (1 hour before food) on Days 1 to 10 plus administration of a single dose of AZD7986 (25 mg) on Day 5 (1 hour before food).
- Itraconazole; OH-itraconazole (a Metabolite of Itraconazole): Participants received Itraconazole (200 mg; oral solution formulation 10 mg/mL) administered twice on Day 1 and then daily on Days 2 to 11 (1 hour before food) plus administration of AZD7986 (25 mg) as a single dose on Day 6 (1 hour before food).
Arm/Group | Verapamil | Itraconazole | OH-itraconazole (a Metabolite of Itraconazole)
Number analyzed (Participants) | 15 | 15 | 15
h*nmol/L | 2178 (44.7) | 18090 (22.6) | 31390 (19.8)

9. Primary Outcome: Assessment of the Tmax of Verapamil, Itraconazole and OH-itraconazole Following Co-administration of AZD7986 With Verapamil or Itraconazole.
Description: To assess the time to reach maximum observed concentration of Verapamil, Itraconazole and OH-itraconazole (a metabolite of itraconazole) following co-administration of AZD7986 with Verapamil or Itraconazole.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Verapamil | Itraconazole | OH-itraconazole (a Metabolite of Itraconazole)
Number analyzed (Participants) | 15 | 15 | 15
hours | 4.00 [1.48 to 12.02] | 1.50 [0.73 to 2.00] | 5.00 [1.00 to 23.93]

ADVERSE EVENTS:
Time Frame: Treatment Period 1: Day -1 up to 96 hours post-dose; Treatment Period 2: Day -1 up to morning of Day 9,; Treatment Period 3: Day -1 up to Day 10 (itraconazole).
Description: An AE is an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. AEs which met the "Definitions of Serious Adverse Event" defined in the clinical study protocol were regarded as SAEs.
Groups:
- Verapamil: Participants received Verapamil
- Itraconazole: Participants received Itraconazole.
- All Subjects: Overall number of participants in the study.
Arm/Group | AZD7986 | AZD7986 + Verapamil | AZD7986 + Itraconazole | Verapamil | Itraconazole | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 7/15 | 5/15 | 3/15 | 6/15 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7986 (N=15) | AZD7986 + Verapamil (N=15) | AZD7986 + Itraconazole (N=15) | Verapamil (N=15) | Itraconazole (N=15) | All Subjects (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 7 (7)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 7 (7)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All of the study information and data collected during the study were considered confidential and the property of AstraZeneca. After completion of the study, the investigator should prepare a joint publication with AstraZeneca. The investigator must undertake not to submit any part of the individual data from this clinical study protocol for publication without prior consent of AstraZeneca at a mutually agreed time.